CLINICAL TRIAL: NCT03730467
Title: Continuation of Breastfeeding After Management of Breast Abscesses by Ultrasound-guided Punctures
Brief Title: Puncture Breast Abscess
Acronym: PONCTABCESEIN
Status: Withdrawn | Type: Observational
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: APHP18022; 2018-A02069-46 (Registry Identifier: ID RCB)
Record Dates: First submitted 2018-11-02; First posted 2018-11-05 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2024-10

CONDITIONS: Breast Abscess
Keywords: Breast feeding; breast abscess; ultrasound-guide; puncture; health
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Phone call to the patient — Phone call to the patient

SUMMARY:
Several breast diseases can complicate breastfeeding : 4% of women develop a mastitis and 1% develop an abscess.

The study deals with cases of breast abscess that have been treated according to a defined protocol (Parisian Perinatal Health Network), by a multidisciplinary team (center of Medical Imaging Duroc) trained in breastfeeding and ultrasound-guided punctures.

The aim of the study is to define the risk factors for the onset of a breast abscess, to evaluate the indications and methods of management of abscess by ultrasound puncture, and to provide arguments motivating the continuation of breastfeeding.

ELIGIBILITY:
Inclusion Criteria:

* Nursing mothers
* Patients referred for breast abscesses during lactation
* Having an abscess confirmed ultrasoundly and indicating a puncture
* Women punctured of an abscess of the breast abscess in the center of Medical Imaging Duroc
* Not opposing the use of them given and to answer the questionnaire on the immediate and medium-term future by telephone
* Women aged > 18 years old
* Women understanding French
* Affiliated to Social Security

Exclusion Criteria:

No

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women punctured for a breast lactant abscess in the center of Medical Imaging Duroc
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2018-09-04 (Actual)

PRIMARY OUTCOMES:
Continuation of breastfeeding | 1 week to 6 months after the puncture
  Phone call to the patient

SECONDARY OUTCOMES:
Etiology of the abscess | 1 week to 6 months after the puncture
  Medical record and phone call to the patient
Adequacy of medical care with the protocol of the Parisian Perinatal Health Network | 1 week to 6 months after the puncture
  Medical record and phone call to the patient
Relationship between puncture breastfeeding continuation | 1 week to 6 months after the puncture
  Medical record and phone call to the patient
Relationship between surgery and weaning | 1 week to 6 months after the puncture
  Medical record and phone call to the patient

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Rigourd, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- AP-HP Hopital Necker Enfants malades, Paris, France